CLINICAL TRIAL: NCT03589404
Title: Investigation of the Effect of Pneumoperitoneum Anterior Abdominal Wall Tissue Oxygenation on Laparoscopic Cholecystectomy
Brief Title: Effect of Pneumoperitoneum Anterior Abdominal Wall Tissue Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Korgün Ökmen, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2018/04-24
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Laparoscopy; Abdominal Wall

STUDY DESIGN:
Intervention Model Description: prospective, cohort,double blind
Masking Description: investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rso2 (Experimental): The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Interventions: Device: rso2

INTERVENTIONS:
Device: rso2 — The regional oxymetry probe will be placed in the abdominal region of the umbilicus in the middle clavicular line before the disease operation begins.
  Other Names: abdominal wall tissue oxygenation

SUMMARY:
During laparoscopic surgery, the abdomen is inflated with carbon dioxide for abdominal imaging and increased intraabdominal pressure affects intraabdominal structures and abdominal wall.

DETAILED DESCRIPTION:
The investigators aimed to investigate the effects of pneumoperitoneum administered during laparoscopic cholecystectomy on abdominal wall oxygenation and postoperative pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were in the American Society of Anesthesiologists (ASA) I-III class
* Underwent laparoscopic cholecystectomy

Exclusion Criteria:

* Previous surgeon surgeon
* Local anesthetic allergy,
* Bleeding is a diathesis disorder
* Mental impairment,
* Allergic to the drugs used,
* Patients who are not reluctant to participate in the study,
* Presence of infection in the block area,
* Patients whose body mass index is over 30

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-15 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
rso2 | perioperative
  The regional oxymetry probe (Medtronic Quick Assist INVOS™ (In-Vivo Optical Spectroscopy) Cerebral/Somatic Oximeter) will be placed in the abdominal region of the umbilicus in the middle clavicular line

SECONDARY OUTCOMES:
Visual Analog Scale | Postoperative 24 hours
  Visual Analog Scale was used for pain.Pain intensity was measured using 0-10 cm visual analogue scale (VAS). (0=no pain, 10=intolerable pain)
analgesic use | Postoperative 24 hours
  analgesic use

CONTACTS AND LOCATIONS:
Overall Officials: Korgün Ökmen, M.D, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No